CLINICAL TRIAL: NCT00756990
Title: Depot Naltrexone Treatment of Opioid Dependent Parolees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 708310
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2019-04-23 (Actual); Status verified 2019-04

CONDITIONS: Opioid Dependence
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single group (Experimental): Depot Naltrexone
  Interventions: Drug: Depot Naltrexone

INTERVENTIONS:
Drug: Depot Naltrexone — 228mg of injectable naltrexone
  Other Names: Depotrex

SUMMARY:
This is an investigation involving the use of a long-acting, injectable form (depot) of naltrexone as a treatment for persons who have a history of opioid dependence, with up to 40 on parole/probation and 20 non-parolees. The test is a pilot study of up to 60 subjects treated with 6 months of depot naltrexone plus Psychosocial Treatment .

DETAILED DESCRIPTION:
This is a two phase study. Phase 1 is complete and phase 2 is not yet recruiting.

ELIGIBILITY:
Inclusion/Exclusion Criteria.

To be eligible to participate, participants must:

* sign an informed consent form;
* be between the ages of 18 and 55;
* have a diagnosis of opioid dependence according to DSM IVTR criteria; and
* be in good general health as determined by complete physical examination and laboratory tests;
* have been assigned to a probation/parole period of at least six months; (except those participants not on parole/probation, see note below); and
* have a negative result for urinary opioids and must self report being at least 3 days opioid free. Participants may have a diagnosis of alcohol dependence so long as they do not have severe alcohol dependence that requires medical supervision for alcohol withdrawal.

Participants with the following characteristics will be excluded from study participation:

* current severe alcohol dependence that requires medical supervision for alcohol withdrawal;
* current psychosis, dementia, mental retardation, or history of schizophrenia;
* significant clinical abnormalities in hematology, chemistry, or urinalysis;
* significant clinical cardiovascular, neurological, hepatic, renal, pulmonary, metabolic, endocrine, or gastrointestinal disorders;
* female subjects who are pregnant or lactating, or female subjects of childbearing potential who are not using birth control (oral contraceptives, barrier (diaphragm or condom) plus spermicide, or levonorgestriel implant);
* subjects who have taken an opioid antagonist within the prior 6 months; and
* current diagnosis of chronic pain disorder.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2005-11; Primary Completion 2009-03 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
UDS results | 6 months

SECONDARY OUTCOMES:
Treatment completion | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Charles O'Brien, MD,PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States